CLINICAL TRIAL: NCT07167654
Title: Effectiveness of a Smartphone Application for Mothers at High Risk for Postpartum Depression: A Randomized Controlled Trial
Brief Title: Smartphone Application to Support Mothers at Risk of Postpartum Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Noor Ali, Principal Investigator, Yarmouk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Yarmouk University
Record Dates: First submitted 2025-08-30; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Depression; Postpartum Depression (PPD)
Keywords: Smartphone Application; psychological interventions; E-Health; postpartum depression; RCT
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention was an Android smartphone application called "Serene Motherhood," which enabled mothers to access evidence-based therapeutic cognitive techniques and health information at any time.
  Interventions: Other: Smartphone Application
- Control group (No Intervention): Control Group who received the routine care for postpartum mothers

INTERVENTIONS:
Other: Smartphone Application — The Intervention: "Serene Motherhood" Application The "Serene Motherhood" application was a newly developed Android-based application created specifically for this study by the research team in collaboration with professional software developers. The content was adapted from authoritative guidelines provided by the American College of Obstetricians and Gynecologists (ACOG), the National Institute for Health and Care Excellence (NICE), the World Health Organization, and the American Psychological Association (APA, 2023; Mota & Bø, 2021; NICE, 2016; WHO, 2022). The application was developed using the research project budget and was provided free of charge to all participants.
  The app aimed to integrate emotional and behavioral strategies, social support, and education for women with symptoms of PPD. The application combines evidence-based therapeutic techniques with user-friendly features supporting daily engagement with the app and self-management. Content and activities were grounded
  Arms: Intervention group

SUMMARY:
Effectiveness of a Smartphone Application for Mothers at High Risk for Postpartum Depression: A Randomized Controlled Trial Abstract

Aim: This study aims to determine the effectiveness of a smartphone application in reducing symptoms of postpartum depression among Jordanian women.

Background: Postpartum depression (PPD) is a serious mental health condition affecting an estimated 14-27% of mothers and negatively impacting infant health. Social support and certain psychological therapies have been shown to reduce depressive symptoms in postpartum women. Smartphone applications may provide a viable means of delivering psychological interventions to mothers experiencing such symptoms.

Method: A randomized controlled trial will be conducted at two maternal and child health clinics in Irbid, Jordan. A total of 295 women will be invited to participate and will be asked to provide sociodemographic data and complete the Edinburgh Postnatal Depression Scale (EPDS) at 6-8 weeks (baseline) and again at 3 months postpartum. Women with a depressive symptom score of ≥13 (n ≈ 79) will be randomly assigned to either the intervention group (n ≈ 58) or the control group (n ≈ 57). The intervention will involve an Android smartphone application called Serene Motherhood, which will enable mothers to access evidence-based cognitive techniques and health information at any time.

DETAILED DESCRIPTION:
Postpartum depression (PPD) is a mental health condition affecting a substantial proportion of mothers during the first year after childbirth. It is characterized by depressed mood, anxiety, feelings of powerlessness or worthlessness, sleep disturbances, and, in some cases, suicidal thoughts. PPD significantly impacts maternal health, leading to physical and psychological difficulties, increased risk of harmful behaviors, social withdrawal, and challenges in performing daily caregiving responsibilities. Infants of affected mothers may experience impaired physical health, irregular sleep patterns, delays in cognitive and emotional development, poor mother-infant bonding, and difficulties initiating and maintaining breastfeeding. These outcomes underscore the importance of early identification and evidence-based interventions.

Psychological interventions, including psychotherapy, support groups, and cognitive-behavioral therapy (CBT), are effective in mitigating PPD symptoms by helping mothers understand their condition, manage negative thoughts, and develop adaptive coping mechanisms. Traditionally, these interventions are delivered face-to-face, providing personal interaction and emotional support. However, multiple barriers, such as socioeconomic limitations, cultural differences, provider bias, time constraints, and limited access in rural or remote areas, often restrict participation in conventional services.

To overcome these barriers, interventions are increasingly delivered remotely through smartphone applications, telephone counseling, and video conferencing platforms. Such approaches offer scalable, flexible, and culturally sensitive options for providing psychological support, particularly to underserved populations. Smartphone applications have shown promise in delivering health education, CBT-based modules, social support, and self-care strategies, with evidence suggesting effectiveness in reducing PPD symptoms in diverse international contexts. Nonetheless, the applicability and outcomes of these interventions in Middle Eastern settings, including Jordan, remain under-investigated.

In Jordan, limited postpartum discharge education and counseling present additional challenges to maternal mental health. Many mothers receive minimal guidance before leaving healthcare facilities, highlighting the need for alternative strategies to support postpartum well-being. At the same time, widespread smartphone access-including in rural communities-offers a feasible platform for delivering interventions that address gaps in education, support, and mental health care.

Given the limited research on smartphone-based interventions for PPD in Arab populations, this study aims to evaluate the effectiveness of a smartphone application specifically designed to support mothers experiencing postpartum depressive symptoms. The study will provide preliminary evidence to inform the potential implementation of scalable digital interventions in Jordan and similar contexts, contributing to improved maternal and infant health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Jordanian women aged 18 to 45 years.
2. Primigravida or multigravida
3. Able to speak and read Arabic
4. Between six and eight weeks postpartum
5. EPDS score of ≥13
6. Access to an Android-compatible smartphone

Exclusion Criteria:

1. Complications during or after childbirth
2. Newborn death or need for special/intensive care
3. Positive response ("yes") to the suicidal ideation item on the EPDS (these participants will be referred to the Prince Basma Outpatient Clinics, Mental Health Department)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — the only eligible self-identified gender is Female.
Enrollment: 79 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-09-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the symptoms of PPD measured by the Edinburgh Postnatal Depression Scale (EPDS) | 12 weeks per participant (from baseline assessment at 6-8 weeks postpartum to follow-up at 3 months postpartum)
  The EPDS is a self-administered questionnaire consisting of ten items, with a total scoring range of 0 to 30 (Cox et al., 1987). Responses are rated on a 4-point scale (0, 1, 2, or 3) according to the severity of symptoms. Items 3, 5, and 10 are reverse-scored (i.e., 3, 2, 1, and 0). The total score is obtained by summing the scores for all ten items, after reversing the coding of negatively worded items, in accordance with the scoring guidelines to ensure consistency.

CONTACTS AND LOCATIONS:
Locations (1):
- Ibn Sina and Hawara Healthcare center, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the sensitive nature of personal and health information related to maternal mental health, which could compromise participant privacy and confidentiality. Only aggregated, de-identified results will be reported.